CLINICAL TRIAL: NCT06728722
Title: Detection of the Changes in Body Composition of Critically Ill Obstetrics by Ultrasound and the Co-relations With Clinical Outcomes; a Prospective Observational Study.
Brief Title: Ultrasound Detection of Body Composition in Critical Care
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU R149/2024
Record Dates: First submitted 2024-10-19; First posted 2024-12-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Muscle Loss; Extracellular Fluid Alteration; Critical Illness; Pregnancy Complications; Gynecologic Disease
Keywords: ultrasound; body composition; critical illness; peripartum and gynecological cases
MeSH Terms: conditions — Muscular Atrophy; Critical Illness; Pregnancy Complications; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- critically ill obstetrics patients , admitted to ICU
  Interventions: Diagnostic Test: ultrasound detection of body composition
- critically ill gynecological cases, admitted to ICU
  Interventions: Diagnostic Test: ultrasound detection of body composition

INTERVENTIONS:
Diagnostic Test: ultrasound detection of body composition — Muscle mass and fat thickness The examiner will use a five-site protocol. The protocol includes the examination of quadriceps on four sides and one bicep will be used The technique is reported by USVALID (Arabella, 2020) GRADING OF QUALITY OF ULTRASOUND SCANS - Muscle quality (fat and fibrotic infiltration) grading for each scan
  1. = Muscle fascia and bone surface visible
  2. = muscle fascia and bone surface still possible to spot
  3. = muscle fascia and bone surface not distinguishable; no evaluation possible
  The FLUID protocol for edema will be done as follows: MEASURING POINTS 36 points, GRADING OF QUALITY: The examiner will use a 5-point scale of ultrasonic subcutaneous edema grade (USEG) to evaluate subcutaneous edema at each site based on echo intensity, tissue transparency, and fluid properties.
  Day zero, day 2 then Every 2 days if extended length.

SUMMARY:
Objective assessment of the Changes in body composition of critically ill patients is very valuable. Ultrasound stands as a solution due to its portability, bedside availability, and radiation-free technology. Those criteria are crucial for critically ill obstetrics and gynecological cases.

DETAILED DESCRIPTION:
Patients with acute/critical illness are particularly vulnerable to muscle loss and fluid shifts, which adversely impact clinical outcomes. Assessment of these parameters in hospital settings is often subjective and imprecise, which creates discrepancies in identification and difficulty in follow-up.

The decrease in muscle mass and/or change in the composition, and fluid overload adversely impact the clinical outcome in critically ill patients and their recovery. There is growing interest in body composition (BC) assessment techniques that can be applied in ICU settings. whole-body BC estimates, and select BC variables show promise as biomarkers of muscle health, nutrition risk, and fluid status. Studies reported that Quadriceps muscle thickness predicted increased morbidity/mortality in ICU patients and has been suggested to be an objective biomarker to determine fitness for aggressive treatment. US measures of muscle loss in the critically ill will aid in the development of appropriate intervention strategies. Alternatively, qualitative muscle evaluation through the measure of echogenicity (using image gray-scale visual analysis) is a sensitive indicator of muscle atrophy. The ultrasound can contribute to assessing necrosis, fatty infiltration, and inflammation in place of invasive muscle biopsy in critically ill patients. Ultrasound offers an important tool for early non-volitional assessment of muscle function in the critically ill.

US characterization of muscle changes would facilitate the development and monitoring of muscle-targeted nutrition and physical therapy interventions. Knowing body muscle and adipose tissue mass is essential in several clinical situations to adapt drug dose to the volume of distribution and to guide nutrition as well as physical therapy. US imaging is a practical method for the prospective assessment of SM (skeletal muscle) changes in response to illness and treatment. Previous ICU studies have focused on measurements of muscle quantity (muscle thickness and CSA) in both the quadriceps, a muscle region known to be rapidly impacted by sarcopenia, and to correlate with ICU survival. Ultrasound has been used primarily as a tool for body composition measurement in clinical nutrition. Although many recent reports have demonstrated that ultrasound could be a useful tool for nutritional assessment and body composition assessment, it is not well incorporated into ICU practice regarding nutritional assessment and follow-up This trial is the first to investigate the role of ultrasound in detecting body composition in critically ill obstetrics and gynecological cases and its correlation with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* females with age 16 with no upper limit
* American Society of Anesthesiologists (ASA) class I, II or III,
* admitted to the obstetrics and Gynecology critical care unit

Exclusion Criteria:

* Patient refusal

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — critically ill pregnant or peripartum or gynecological critical illness
Study Population: Critically ill women whether pregnant, peripartum, postoperative, or admitted for any critical illness.
Sampling Method: Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
change in body composition-muscular element | on the day of admission , repeated every 2 days till death or discharge which come first, assessed up to 20 days from admission
  Decreased muscle thickness measured by mm or change in quality by visual frey-white detection by ultrasound. The grading for each scan
  1. = Muscle fascia and bone surface visible
  2. = muscle fascia and bone surface still possible to spot
  3. = muscle fascia and bone surface not distinguishable; no evaluation possible
change in body composition-fat element | on the day of admission , repeated every 2 days till death or discharge which come first, assessed up to 20 days from admission.
  change in thickness of subcutaneous fat measured in mm.
change in body composition-extreacellular oedema element | on the day of admission , repeated every 2 days till death or discharge which come first .
  The examiner will use a 5-point scale of ultrasonic subcutaneous edema grade (USEG) to evaluate subcutaneous edema at each site based on echo intensity, tissue transparency, and fluid properties.
  the total Degree of edema measurement is: The final ultrasonic subcutaneous edema score (USES) will be calculated by adding scores from 36 subcutaneous sites (0-144). Each regional score will be estimated by summing the site scores of the hands (0-8), arms (0-16), thoracic wall (0-32), abdominal wall (0-32), thigh (0-24), calves (0-24), and feet (0-8). The total regional score will be divided by the number of sites in each region to the average score (0-4). the lower the score = the lower level of edema.

SECONDARY OUTCOMES:
co-relation of the change of any elements of body composition with poor outcomes suchs such as death, need for ventilatory or circulatory support or increase the length of stay in icu. | from occurence of change in body composition till the poor outcome. till discharge from icu or death which come first, assessed till 20 days from admission
  Positive co-relation or negative correlation between both. That will be measured by the frequency of occurrence of poor clinical outcomes-mortality cardiorespiratory support or prolonged length of stay- in patients with positive change in any element (muscular-fat-extracellular edema).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: it will be available after completion and acceptance from a peer reviewed journal and upon reasonable request
Access Criteria: upon reasonable request from one of the authors.

REFERENCES:
- [Background] Gursoy C, Alkan A, Kaya Cubuk E, Karci E, Yilmaz HO, Cakir T. Rectus abdominis and rectus femoris muscle thickness in determining nutritional risk in critically ill patients: a prospective cohort study in Turkey. BMJ Open. 2023 Mar 30;13(3):e071796. doi: 10.1136/bmjopen-2023-071796. PMID 36997242
- [Background] Ponti F, De Cinque A, Fazio N, Napoli A, Guglielmi G, Bazzocchi A. Ultrasound imaging, a stethoscope for body composition assessment. Quant Imaging Med Surg. 2020 Aug;10(8):1699-1722. doi: 10.21037/qims-19-1048. PMID 32742962
- [Background] Zhang W, Gu Y, Zhao Y, Lian J, Zeng Q, Wang X, Wu J, Gu Q; Chinese Critical Care Ultrasound Study Group (CCUSG). Focused liquid ultrasonography in dropsy protocol for quantitative assessment of subcutaneous edema. Crit Care. 2023 Mar 18;27(1):114. doi: 10.1186/s13054-023-04403-y. PMID 36934293